CLINICAL TRIAL: NCT04136951
Title: Improving Patient Prioritization During Hospital-homecare Transition: A Mixed Methods Study of a Clinical Decision Support Tool
Brief Title: Improving Patient Prioritization During Hospital-homecare Transition
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Visiting Nurse Service of New York (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maxim Topaz, Associate Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AAAS7265; 1R01NR018831-01 (NIH)
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2; Congestive Heart Failure; Obstructive Pulmonary Disease; Dyspnea; Renal Failure
Keywords: home health; clinical decisions support; care transitions; patient prioritization; health informatics; home care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Lung Diseases, Obstructive; Dyspnea; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: To examine the study aims, the researchers are using an embedded mixed methods study design. The researchers will conduct pre- and post intervention trial of clinical decision support tool PREVENT's integration into clinical practice using homecare admissions from two New York City urban hospitals serving diverse racial and ethnic population. Quantitative methods, including logistic regression and survival analysis with propensity score matching, will be used to evaluate the effects of the tool on process and patient outcomes. Qualitative methods will be used to match the quantitative questions and provide an in depth insight into homecare admission processes using think-aloud simulations and interviews with homecare admission staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental phase (Experimental): The PREVENT recommendation about patient homecare priority will be shared in homecare referral communication with the homecare intake coordinators. Homecare intake coordinators will be instructed to prioritize high risk patients for care.
  Interventions: Other: PREVENT clinical decision support

INTERVENTIONS:
Other: PREVENT clinical decision support — PREVENT clinical decision support tool consideres five patient risk factors as significant predictors of patient's priority for the first homecare nursing visit: (a) Presence of wounds (either surgical or pressure ulcers); (b) a documented comorbid condition of depression; (c) need for assistive equipment, assistive person, or both for toileting; (d) number of medications; and (e) number of comorbid conditions. Each risk factor was assigned a specific score based on the logistic regression weights. For instance, for a wound (e.g., pressure ulcer, vascular ulcer), the patient received a score of 15 points. For each additional co-morbid condition, one point was added to the final score. Summing the scores for the factors generated a cumulative score. The optimal cut-off point was established based on the regression model performance statistics, indicating that patients with a score greater than 26 points are a high priority for the first nursing visit.

SUMMARY:
This research work is focused on building and evaluating one of the first evidence-based clinical decision support tools for homecare in the United States. The results of this study have the potential to standardize and individualize nursing decision making using cutting-edge technology and to improve patient outcomes in the homecare setting.

DETAILED DESCRIPTION:
Each year, more than 5 million patients are admitted to the approximately 12,000 homecare agencies across the United States. About 20% of homecare patients are rehospitalized during the homecare episode, with as many as 68% of these rehospitalizations occurring within the first two weeks of services. A significant portion of these rehospitalizations may be prevented by timely and appropriately targeted allocation of homecare services. The first homecare nursing visit is one of the most critical steps of the homecare episode. This visit includes an examination of the home environment, a discussion regarding whether a caregiver is present, an assessment of the patient's capacity for self-care, and medication reconciliation. A unique care plan is created based on this evaluation of the patient's needs. Hence, appropriate timing of the first visit is crucial, especially for patients with urgent healthcare needs. However, nurses often have very limited and inaccurate information about incoming patients and patient priority decisions vary significantly between nurses.

The investigators developed an innovative decision support tool called "Priority for the First Nursing Visit Tool" (PREVENT) to assist nurses in prioritizing patients in need of immediate first homecare nursing visits. In a recent efficacy pilot study of PREVENT, high-risk patients received their first homecare nursing visit a half day sooner as compared to the control group, and 60-day rehospitalizations decreased by almost half as compared to the control group. The proposed study assembles a strong interdisciplinary team of experts in health informatics, nursing, homecare, and sociotechnical disciplines to evaluate PREVENT in a pre-post intervention effectiveness study. Specifically, the study aims are: Aim 1) Evaluate the effectiveness of the PREVENT tool on process and patient outcomes. Using survival analysis and logistic regression with propensity score matching the researchers will test the following hypotheses: Compared to not using the tool in the pre-intervention phase, when homecare clinicians use the PREVENT tool, high risk patients in the intervention phase will: a) receive more timely first homecare visits and b) have decreased incidence of rehospitalization and have decreased emergency department (ED) use within 60 days. Aim 2) Explore PREVENT's reach and adoption by the homecare admission staff and describe the tool's implementation during homecare admission. Aim 2 will be assessed using mixed methods including homecare admission staff interviews, think-aloud simulations, and analysis of staffing and other relevant data.

This innovative study addresses several National Institute of Nursing Research strategic priorities, such as promoting innovation and using technology to improve health. Mixed methods will enable us to gain in-depth understanding of the complex socio-technological aspects of hospital-homecare transition.

ELIGIBILITY:
Aim 1:

Inclusion criteria:

1. being a patient of either NewYork-Presbyterian (NYP)/Columbia University Irving Medical Center or NewYork-Presbyterian Allen Hospital;
2. being referred to Visiting Nurse Services of New York (VNSNY) homecare services
3. 18 years old or older.

Exclusion criteria:

All other patients are going to be excluded.

Aim 2 :

Inclusion criteria:

1. working as an admission staff for VNSNY
2. 18 years old or older.

Exclusion criteria:

All other staff members are going to be excluded.

For both study aims, there will be no exclusion based on sex, race, or ethnic group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1915 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Topaz, PhD, Principal Investigator — Associate Professor of Nursing at CUMC
Locations (2):
- United States (2):
  - Columbia University School of Nursing, New York, New York
  - Visiting Nurse Service of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No
No sharing planned

REFERENCES:
- [Result] Topaz M, Trifilio M, Maloney D, Bar-Bachar O, Bowles KH. Improving patient prioritization during hospital-homecare transition: A pilot study of a clinical decision support tool. Res Nurs Health. 2018 Oct;41(5):440-447. doi: 10.1002/nur.21907. Epub 2018 Sep 11. PMID 30203417
- [Derived] Zolnoori M, McDonald MV, Barron Y, Cato K, Sockolow P, Sridharan S, Onorato N, Bowles K, Topaz M. Improving Patient Prioritization During Hospital-Homecare Transition: Protocol for a Mixed Methods Study of a Clinical Decision Support Tool Implementation. JMIR Res Protoc. 2021 Jan 22;10(1):e20184. doi: 10.2196/20184. PMID 33480855

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: home healthcare admissions
Groups:
- PREVENT: Data will be calculated from patients referred to the Visiting Nurse Service of New York from the 2 hospitals (NewYork-Presbyterian Hospital/Columbia University Irving Medical Center and NYP Allen Hospital) in a 3 month period during the preintervention phase (scores not shared) and a 3 month intervention phase (scores shared).
Period: Pre-intervention Phase (3 Months)
Arm/Group | PREVENT
Started | 1915; 1048 home healthcare admissions
Completed | 1915; 1048 home healthcare admissions
Not Completed | 0; 0 home healthcare admissions
Period: Intervention Phase (3 Months)
Arm/Group | PREVENT
Started | 1915; 970 home healthcare admissions
Completed | 1915; 970 home healthcare admissions
Not Completed | 0; 0 home healthcare admissions

BASELINE CHARACTERISTICS:
Arm/Group | PREVENT
Number analyzed (Participants) | 1915
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1915
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1113
  Male | 802
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 375
  Hispanic | 923
  White | 492
  Other | 125
  Unknown/Not reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1915

OUTCOME MEASURES:

1. Primary Outcome: Number of Rehospitalizations Within 60 Days After Hospital Discharge
Description: To learn if using PREVENT tool results in decreased incidence of rehospitalization [defined as recurrent hospital admission within 60 days from hospital discharge]
Time Frame: Up to 60 days after hospital discharge
Measure: Number; unit: rehospitalizations
Arm/Group | PREVENT
Number analyzed (Participants) | 1915
rehospitalizations | 807

2. Other Pre Specified Outcome: System Usability Scale (SUS) Score
Description: Nurses' usability perception of the clinical decision support tool (PREVENT) will be assessed by using the System Usability Scale (SUS). The SUS is a 10 item questionnaire, each with a five-point Likert scale, allowing users to rate their agreement or disagreement. The SUS score is calculated by converting the raw scores from the Likert scale and then multiplying the sum by 2.5, resulting in a score between 0 and 100, where a higher score indicates greater perceived usability.
Time Frame: 30-60 days after clinical decision support tool (PREVENT) implementation
Population: Due to operational constraints during implementation, the SUS survey was not administered to nursing staff.
Arm/Group | PREVENT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 60 days following each home healthcare admission
Description: Adverse event data was collected through retrospective electronic health records review
Arm/Group | PREVENT
All-Cause Mortality (participants affected / at risk) | 0/1915
Serious Adverse Events (participants affected / at risk) | 0/1915
Other Adverse Events (participants affected / at risk) | 0/1915

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04136951/Prot_SAP_000.pdf